CLINICAL TRIAL: NCT00796705
Title: Switching Anti-TNF-alpha Agents in Patients With RA With An Inadequate Response to TNF-alpha Inhibition
Brief Title: Switching Anti-TNF-Alpha Agents in Rheumatoid Arthritis (RA)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ARA05
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Results first posted 2012-08-13 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adalimumab / Adalimumab Placebo (Experimental): 1 sub-cutaneous (SQ) injection of adalimumab or 1 SQ injection of placebo will be given in a blinded and alternating fashion for a total of 12 weeks
  Interventions: Drug: Adalimumab; Drug: Adalimumab placebo
- Etanercept (Experimental): Participants will receive 1 SQ injection of etanercept each week for 12 weeks
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Adalimumab — 40 mg injection of adalimumab administered subcutaneously
  Other Names: Humira
  Arms: Adalimumab / Adalimumab Placebo
Drug: Adalimumab placebo — 1.0 ml .9% saline placebo administered subcutaneously
  Other Names: Humira placebo
  Arms: Adalimumab / Adalimumab Placebo
Drug: Etanercept — 50 mg dimeric fusion protein administered subcutaneously
  Other Names: Enbrel
  Arms: Etanercept

SUMMARY:
Rheumatoid Arthritis (RA) is a systemic inflammatory autoimmune disorder that leads to inflammation and progressive joint damage affecting 2.5 million people in the United States. The primary purpose of this study is to determine the effectiveness of switching to an alternative Tumor Necrosis Factor (TNF) alpha inhibitor in comparison to continuing treatment with an existing TNF-alpha inhibitor in adults suffering from RA in a setting of inadequate clinical response to etanercept or adalimumab.

DETAILED DESCRIPTION:
Over the past 10 years, advancements in biotechnology have revolutionized Rheumatoid Arthritis (RA) therapeutics with biologically-derived immunomodulating compounds. Tumor Necrosis Factor (TNF) alpha inhibitors constitute the largest class of these new biologic therapies. The purpose of this study is to determine the effectiveness of switching to an alternative TNF-alpha inhibitor in comparison to continuing treatment with an existing TNF-alpha inhibitor in adults suffering from RA who have had inadequate clinical response to the study drugs etanercept and adalimumab.

This study will last approximately 16 weeks. Participants will be randomized into two arms and receive injections once per week for 12 weeks. Participants in the adalimumab arm will receive alternating subcutaneous adalimumab and adalimumab placebo injections. Participants in the etanercept arm will receive subcutaneous etanercept injections.

This study consists of thirteen study visits after randomization. Study visits will occur on a weekly basis for 12 weeks prior to a follow-up visit at Week 16. A vital signs measurement and adverse event assessment will occur at each visit. A physical exam, assessment of tender and swollen joints, medication assessment, and blood collection will occur at Weeks 4, 8, 12, and 16.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis
* Current treatment with either etanercept or adalimumab for at least 12 weeks prior to randomization
* Disease Activity Score (DAS) C-reactive Protein (CRP) 28 ≥ 4.4
* Treatment with concomitant Disease-Modifying Anti-Rheumatic Drugs (DMARDs) is permitted but not required as described below:

  1. Methotrexate - maximum dose of 25 mg per os (PO), intra-muscular (IM), or SQ weekly.
  2. Leflunomide - maximum dose of 20 mg PO daily.
  3. Sulfasalazine - maximum dose of 1,500 mg PO twice daily.
  4. Hydroxychloroquine - maximum dose of 400 mg PO daily.
* If taking DMARD(s), subjects must be on stable doses for at least 12 weeks prior to randomization.
* If treated with prednisone (or equivalent corticosteroid), on a stable dose of <= 10 mg/day for 28 days prior to randomization.
* Agree to use appropriate form of contraception. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Diagnosis of another autoimmune disease likely to require immunosuppression. More information on this criterion can be found in the protocol.
* Failing treatment with etanercept if previously treated with adalimumab
* Failing treatment with adalimumab if previously treated with etanercept
* Intraarticular injection within 4 weeks prior to randomization
* Concomitant use of DMARDs other than those described in Inclusion Criteria within 12 weeks of randomization.
* Concurrent use of any biologic agent other than etanercept or adalimumab
* Concomitant immunosuppressive therapy other than the Disease-Modifying Anti-Rheumatic Drugs (DMARDs), non-steroidal anti-inflammatory drugs (NSAIDs), or corticosteroids specified in the protocol
* Presence of open leg ulcers
* Chronic or persistent infection that may be worsened by immunosuppressive treatment. More information on this criterion can be found in the protocol.
* Active infection or severe infections requiring hospitalization or treatment with intravenous antibiotics, antivirals, or antifungals within 30 days prior to randomization
* History of positive Purified Protein Derivative (PPD) or chest x-ray findings indicative of prior tuberculosis infection
* Any medical condition or treatment that, in the opinion of the investigator, would put the subject at risk by participation in the study
* History of malignancy. More information on this criterion can be found in the protocol.
* Certain abnormal laboratory values. More information on this criterion can be found in the protocol.
* Investigational biological or chemical agents within 4 weeks prior to randomization.
* History of drug or alcohol abuse within a year prior to randomization
* Treatment with natalizumab, rituximab, or another B-cell depleting therapy within a year prior to randomization
* Treatment with infliximab, abatacept, tocilizumab, golimumab, or certolizumab pegol within 12 weeks prior to randomization.
* Known allergy or hypersensitivity to study products
* Any psychiatric disorder that prevents the participant from providing informed consent
* Inability to follow protocol instructions
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Moreland, MD, Study Chair — University of Pittsburgh; Mark Genovese, MD, Study Chair — Stanford University
Locations (16):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Tampa Medical Group, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Justus Fiechtner, MD, PC, Lansing, Michigan
  - Feinstein Institute for Medical Research NS-LIJ, Manhassett, New York
  - University of Rochester, Rochester, New York
  - Carolina Bone and Joint, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor Research Institute, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Villeneuve E, Haraoui B. To switch or to change class-the biologic dilemma in rheumatoid arthritis. Nat Rev Rheumatol. 2010 May;6(5):301-5. doi: 10.1038/nrrheum.2010.45. Epub 2010 Apr 13. PMID 20386564
- [Background] Rubbert-Roth A, Finckh A. Treatment options in patients with rheumatoid arthritis failing initial TNF inhibitor therapy: a critical review. Arthritis Res Ther. 2009;11 Suppl 1(Suppl 1):S1. doi: 10.1186/ar2666. Epub 2009 Apr 6. PMID 19368701
- [Background] van Gestel AM, Haagsma CJ, van Riel PL. Validation of rheumatoid arthritis improvement criteria that include simplified joint counts. Arthritis Rheum. 1998 Oct;41(10):1845-50. doi: 10.1002/1529-0131(199810)41:103.0.CO;2-K. PMID 9778226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred between November 2008 and November 2010 at 16 sites located in the United States. All sites utilized a rheumatology clinic and outside referrals for recruitment.
Pre-assignment Details: Each subject signed an informed consent prior to undergoing any screening procedures. At the screening visit, subjects underwent procedures to establish inclusion/exclusion criteria.
Groups:
- Non-Switcher/Adalimumab Alternating With Placebo: Participants defined as adalimumab failures [1] at screening who were randomized to remain on adalimumab (one 40 milligram [mg] subcutaneous [SQ] injection) alternating with adalimumab placebo (1.0 millilitre [mL] SQ injection of normal saline 0.9%) once weekly for a total of 12 weeks in a blinded (masked) fashion.
  [1] Adalimumab failures: participants with rheumatoid arthritis [RA] on adalimumab treatment for at least 12 weeks prior to treatment randomization that experienced inadequate clinical response to adalimumab.
- Non-Switcher/Etanercept: Participants defined as etanercept failures [1] at screening who were randomized to receive etanercept (one 50 mg subcutaneous injection) once weekly for a total of 12 weeks in a blinded (masked) fashion.
  [1] Etanercept failures: participants with rheumatoid arthritis [RA] on etanercept treatment for at least 12 weeks prior to randomization that experienced inadequate clinical response to etanercept.
- Switcher/Adalimumab to Etanercept: Participants defined as adalimumab failures [1] at screening who were randomized to switch from adalimumab to etanercept (one 50 mg subcutaneous injection) once weekly for a total of 12 weeks in a blinded (masked) treatment fashion.
  [1] Adalimumab failures: participants with rheumatoid arthritis [RA] on adalimumab treatment for at least 12 weeks prior to treatment randomization that experienced inadequate clinical response to adalimumab.
- Switcher/Etanercept to Adalimumab Alternating With Placebo: Participants defined as etanercept failures [1] at screening who were randomized to switch from etanercept to adalimumab (one 40 mg subcutaneous [SQ] injection) alternating with adalimumab placebo (1.0 mL SQ injection of normal saline 0.9%) once weekly for a total of 12 weeks in a blinded (masked) fashion.
  [1] Etanercept failures: participants with rheumatoid arthritis [RA] on etanercept treatment for at least 12 weeks prior to randomization that experienced inadequate clinical response to etanercept.
Period: Overall Study
Arm/Group | Non-Switcher/Adalimumab Alternating With Placebo | Non-Switcher/Etanercept | Switcher/Adalimumab to Etanercept | Switcher/Etanercept to Adalimumab Alternating With Placebo
Started | 3 | 4 | 4 | 2
Completed | 3 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Switcher/Adalimumab to Etanercept: Participants defined as adalimumab failures [1]at screening who were randomized to switch from adalimumab to etanercept (one 50 mg subcutaneous injection) once weekly for a total of 12 weeks in a blinded (masked) treatment fashion.
  [1] Adalimumab failures: participants with rheumatoid arthritis [RA] on adalimumab treatment for at least 12 weeks prior to treatment randomization that experienced inadequate clinical response to adalimumab.
- Total: Total of all reporting groups
Arm/Group | Non-Switcher/Adalimumab Alternating With Placebo | Non-Switcher/Etanercept | Switcher/Adalimumab to Etanercept | Switcher/Etanercept to Adalimumab Alternating With Placebo | Total
Number analyzed (Participants) | 3 | 4 | 4 | 2 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 4 | 2 | 11
  >=65 years | 0 | 2 | 0 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (4.0) | 65 (9.4) | 39 (13.7) | 60 (6.4) | 53 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 2 | 13
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 4 | 2 | 13
Disease Activity Score Using C-reactive Protein (DAS28[CRP]) [Mean (Standard Deviation); unit: Scores on a scale] — The DAS28 is: a score on a scale (0 to 10) indicating current activity of rheumatoid arthritis (>5.1=high disease activity; <=3.2=low disease activity; <2.6=remission); a continuous variable which is a composite of 4 variables(the number of tender joints out of 28, the number of swollen joints out of 28 joints, serum C-reactive protein in mg/L (CRP) and subject assessment of disease activity measure on a visual analogue scale (VAS) of 100 mm).
  Scores on a scale | 5.6 (0.66) | 5.4 (0.44) | 4.8 (0.62) | 5.3 (0.19) | 5.3 (0.56)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Disease Activity Score Using C-reactive Protein (DAS28[CRP]) From Baseline to Week 12 in Non-Switchers Versus Switchers.
Description: The DAS28 is a score on a scale (0 to 10) indicating current activity of rheumatoid arthritis (>5.1=high disease activity; <=3.2=low disease activity; <2.6=remission); a continuous variable which is a composite of 4 variables(the number of tender joints out of 28, the number of swollen joints out of 28 joints, serum C-reactive protein in mg/L (CRP) and subject assessment of disease activity measure on a visual analogue scale (VAS) of 100 mm).
Time Frame: Baseline, Week 12
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Non-Switcher/ Adalimumab or Etanercept: Participants defined as adalimumab failures [1] at screening who were randomized to remain on adalimumab (one 40 milligram [mg] subcutaneous [SQ] injection) alternating with adalimumab placebo (1.0 millilitre [mL] SQ injection of normal saline 0.9%) once weekly for a total of 12 weeks in a blinded (masked) fashion and participants defined as etanercept failures [2] at screening who were randomized to receive etanercept (one 50 mg SQ injection) once weekly for a total of 12 weeks in a blinded (masked) fashion.
  1. Adalimumab failures: participants with rheumatoid arthritis [RA] on adalimumab treatment for at least 12 weeks prior to treatment randomization that experienced inadequate clinical response to adalimumab.
  2. Etanercept failures: participants with rheumatoid arthritis [RA] on etanercept treatment for at least 12 weeks prior to randomization that experienced inadequate clinical response to etanercept.
- Switcher/ Adalimumab to Etanercept or Etanercept to Adalimuma: Participants defined as adalimumab failures [1]at screening who were randomized to switch from adalimumab to etanercept (one 50 mg SQ injection) once weekly for a total of 12 weeks in a blinded (masked) treatment fashion and participants defined as etanercept failures [2] at screening who were randomized to switch from etanercept to adalimumab (one 40 mg SQ injection) alternating with adalimumab placebo (1.0 mL SQ injection of normal saline 0.9%) once weekly for a total of 12 weeks in a blinded (masked) fashion.
  1. Adalimumab failures: participants with rheumatoid arthritis [RA] on adalimumab treatment for at least 12 weeks prior to treatment randomization that experienced inadequate clinical response to adalimumab.
  2. Etanercept failures: participants with rheumatoid arthritis [RA] on etanercept treatment for at least 12 weeks prior to randomization that experienced inadequate clinical response to etanercept.
Arm/Group | Non-Switcher/ Adalimumab or Etanercept | Switcher/ Adalimumab to Etanercept or Etanercept to Adalimuma
Number analyzed (Participants) | 7 | 6
Scores on a scale | -1.4 (0.90) | -1.7 (1.09)

2. Primary Outcome: Change in the Disease Activity Score Using C-reactive Protein (DAS28[CRP]) From Baseline to Week 12.
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-Switcher/Adalimumab Alternating With Placebo | Non-Switcher/Etanercept | Switcher/Adalimumab to Etanercept | Switcher/Etanercept to Adalimumab Alternating With Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 2
Scores on a scale | -2.0 (0.22) | -0.9 (0.92) | -1.7 (0.94) | -1.5 (1.81)

3. Secondary Outcome: Participants With a Disease Activity Score Using C-reactive Protein (DAS28[CRP]) Value <= 3.2 (Low Disease Activity) at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Non-Switcher/Adalimumab Alternating With Placebo | Non-Switcher/Etanercept | Switcher/Adalimumab to Etanercept | Switcher/Etanercept to Adalimumab Alternating With Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 2
participants | 1 | 1 | 2 | 1

4. Secondary Outcome: Participants With a Disease Activity Score Using C-reactive Protein (DAS28[CRP]) Value < 2.6 (Remission) at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Non-Switcher/Adalimumab Alternating With Placebo | Non-Switcher/Etanercept | Switcher/Adalimumab to Etanercept | Switcher/Etanercept to Adalimumab Alternating With Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 2
participants | 0 | 0 | 1 | 1

5. Secondary Outcome: Participants With a Decrease in Disease Activity Score Using C-reactive Protein (DAS28[CRP]) Value of >1.2 From Baseline to Week 12 (European League Against Rheumatism (EULAR) Definition of a Moderate Response)
Description: The EULAR definition of a Moderate Response is a decrease from baseline in the DAS28[CRP] value of ≥ 1.2.
Time Frame: Baseline, Week 12
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Non-Switcher/Adalimumab Alternating With Placebo | Non-Switcher/Etanercept | Switcher/Adalimumab to Etanercept | Switcher/Etanercept to Adalimumab Alternating With Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 2
participants | 3 | 1 | 2 | 1

6. Secondary Outcome: Participants With an ACR 20 Response at Week 12
Description: The American College of Rheumatology (ACR) 20 Responder Index is defined as someone who achieved at least 20% improvement in the tender and swollen 28-joint count, and 20% improvement in at least three of the following 5 measures:
  * Patient's pain assessment (Visual Analogue Scale (VAS) 100 mm)
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (CRP)
Time Frame: Week 12
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Non-Switcher/Adalimumab Alternating With Placebo | Non-Switcher/Etanercept | Switcher/Adalimumab to Etanercept | Switcher/Etanercept to Adalimumab Alternating With Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 2
participants | 3 | 2 | 3 | 1

7. Secondary Outcome: Participants With an ACR 50 Response at Week 12
Description: The American College of Rheumatology (ACR) 50 Responder Index is defined as someone who achieved at least 50% improvement in the tender and swollen 28-joint count, and 50% improvement in at least three of the following 5 measures:
  * Patient's pain assessment (Visual Analogue Scale (VAS) 100 mm)
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (CRP)
Time Frame: Week 12
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Non-Switcher/Adalimumab Alternating With Placebo | Non-Switcher/Etanercept | Switcher/Adalimumab to Etanercept | Switcher/Etanercept to Adalimumab Alternating With Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 2
participants | 2 | 0 | 1 | 0

8. Secondary Outcome: Participants With an ACR 70 Response at Week 12
Description: The American College of Rheumatology (ACR) 70 Responder Index is defined as someone who achieved at least 70% improvement in the tender and swollen 28- joint count, and 70% improvement in at least three of the following the following 5 measures:
  * Patient's pain assessment (Visual Analogue Scale (VAS) 100 mm)
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (CRP)
Time Frame: Week 12
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Non-Switcher/Adalimumab Alternating With Placebo | Non-Switcher/Etanercept | Switcher/Adalimumab to Etanercept | Switcher/Etanercept to Adalimumab Alternating With Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 2
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Non-Switcher/Adalimumab: Subjects failing Adalimumab at screening who were randomized to remain on Adalimumab
- Non-Switcher/Etanercept: Subjects failing Etanercept at screening who were randomized to remain on Etanercept
- Switcher/Adalimumab to Etanercept: Subjects failing Adalimumab at screening who were randomized to switch to Etanercept
- Switcher/Etanercept to Adalimumab: Subjects failing Etanercept at screening who were randomized to switch to Adalimumab
Arm/Group | Non-Switcher/Adalimumab | Non-Switcher/Etanercept | Switcher/Adalimumab to Etanercept | Switcher/Etanercept to Adalimumab
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 4/4 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Switcher/Adalimumab (N=3) | Non-Switcher/Etanercept (N=4) | Switcher/Adalimumab to Etanercept (N=4) | Switcher/Etanercept to Adalimumab (N=2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site irritation (General disorders) | 0 (0) | 2 (6) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 2 (7) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallop rhythm present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study terminated early due to recruitment feasibility issues. Thirteen subjects were enrolled and received treatment. No mechanistic analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No